CLINICAL TRIAL: NCT02144571
Title: SCCDCN-II: Research Project (Breast Cancer)
Brief Title: Sistas Inspiring Sistas Through Activity and Support
Acronym: SISTAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, James hebert, Dr. Jame Hebert, University of South Carolina
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00008713
Record Dates: First submitted 2014-05-12; First posted 2014-05-22 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Prevention Harmful Effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle (Experimental): Diet and physical activity intervention group. Measurements taken at baseline, 12 weeks and 1 year.
  Interventions: Behavioral: Lifestyle
- Wait-list control (No Intervention): No-treatment control group. Measurements taken at baseline, 12 weeks and 1 year. People in the control condition can elect to take the intervention after 1 year.

INTERVENTIONS:
Behavioral: Lifestyle — Participants are consented and randomized into the intervention group or delayed intervention group(intervention offered one year later). Participants in intervention group attend 12 weekly sessions and 9 monthly sessions. All participants attend 3 clinics in which we collect data, measurements and blood samples. These clinics occur at baseline, 12 weeks and one year.
  Other Names: SISTAS
  Arms: Lifestyle

SUMMARY:
It is known that diet and physical affect a variety of disease-related endpoints and overall health status in general. The investigators also know that dietary and PA intervention effects are difficult for individuals to maintain. By contrast, the investigators have some evidence that group-based and family-centered, multi-component interventions are more effective in terms of creating large changes in diet-related outcomes. Using a group-randomized, controlled design, the overall goal of this project is to reduce breast cancer-related health disparities in a high-risk community, by achieving these Primary Aims,to conduct a regionally-based community-designed dietary and physical activity behavioral controlled trial among AA women,to test the effectiveness of the community-designed, family-based dietary and physical activity behavioral intervention on modifying biomarkers of inflammation and to test the effectiveness of the community-designed, family-based dietary and physical activity behavioral intervention on decreasing breast density

DETAILED DESCRIPTION:
AAs in South Carolina bear an unequal burden of cancer incidence and mortality compared to their European American counterparts. The Research Program (RP) is committed to investigating and eliminating this burden through the careful conduct of research studies in partnership with their AA community partners. The overall aim of the RP is to support the SCCDCN-II in its mission to reduce, and ultimately eliminate, cancer health disparities using a community-based participatory research (CBPR) approach to design and conduct research projects in AA communities in South Carolina. The goals of the research program are to: support the SCCDCN by serving as a research liaison/consultant for all community-based activities; foster and support meaningful partnerships between academic researchers and community leaders and representatives; conduct a two-arm physical activity and dietary intervention trial for breast cancer prevention among African-American women in the investigators target communities of faith; conduct a pilot study to determine African-American men's and women's knowledge about prostate cancer screening and their knowledge and attitudes regarding participation in prostate cancer research, including National Cancer Institute (NCI) sponsored clinical trials; support additional research in cancer disparities through a Pilot Study post-transition year and to develop and implement an SCCDCN-II internal pilot grants program in years 4 and 5; and partner with community representatives to disseminate program findings and to work with colleagues in the AC, and Community Outreach and Training Programs to develop community capacity aimed at sustaining programs to improve health The two-arm intervention trial will be aimed at testing the effectiveness of a community-designed, family-based dietary and PA behavioral intervention on modifying biomarkers of inflammation and decreasing breast density with a randomized controlled design. The prostate cancer pilot will be aimed at assessing current knowledge and attitudes regarding prostate cancer prevention and screening, and participation in prostate cancer research; changes in knowledge and attitudes about research participation following a pilot education program; and culturally appropriate strategies for promoting cancer research among AAs in a faith-based community. All activities of the research program will be conducted in partnership with identified SCCDCN II community partners, the State Baptist YWA of the Women's BEMC, SCPHCA, CCBHSN, and Insights Consulting. It is anticipated that research activities will be conducted in all 5 years of the granting period with opportunities for research partnerships in all State Baptist YWA regions throughout the state.

ELIGIBILITY:
Inclusion Criteria:

* 30 years of age or older
* African American
* BMI 30 or<
* Willing to be randomized,

Exclusion Criteria:

* History of cancer
* Inflammatory-related conditions
* Unstable hormones replacement treatment

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2010-11; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Inflammatory Response | Baseline, 12 weeks and 12 months
  This will entail examining changes in the inflammatory index derived from dietary self-report and self-reported physical activity and blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Swann Arp-Adams, Ph.D, Study Director — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request using our data request form and with data committee approval. We will allow the data to be shared after publication of our two primary outcome manuscripts.